CLINICAL TRIAL: NCT03973203
Title: The Effect of Niacin Supplementation on Systemic Nicotinamide Adenine Dinucleotide (NAD+) Metabolism, Physiology and Muscle Performance in Healthy Controls and Mitochondrial Myopathy Patients
Brief Title: Niacin Supplementation in Healthy Controls and Mitochondrial Myopathy Patients
Acronym: NiaMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other); Institute for Molecular Medicine (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, Anu Wartiovaara, Academy Professor, Professor of Clinical Molecular Medicine, University of Helsinki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NiaMIT_0001
Record Dates: First submitted 2019-05-24; First posted 2019-06-04 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Mitochondrial Myopathies
Keywords: vitamin B3; niacin; mitochondrial myopathy; mitochondria; muscle; muscle strength; NAD+ precursor; NAD+; NAD-booster
MeSH Terms: conditions — Mitochondrial Myopathies | interventions — Niacin

STUDY DESIGN:
Intervention Model Description: All participants (healthy controls and mitochondrial myopathy patients) receive orally administered a slow-released form of niacin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niacin in controls (Experimental): The arm includes healthy controls supplemented with niacin.
  Interventions: Dietary Supplement: Niacin
- Niacin in mitochondrial myopathy patients (Experimental): The arm includes mitochondrial myopathy patients supplemented with niacin.
  Interventions: Dietary Supplement: Niacin

INTERVENTIONS:
Dietary Supplement: Niacin — The dose for a slow-released form of niacin will be 750-1000 mg/day. The daily niacin dose, 250 mg/day, is gradually escalated by 250 mg/month so that the full dose is reached after 3 months. The intervention time with the full niacin dose is 1 and 7 months for controls and patients, respectively, and subsequently total intervention time 4 and 10 months, respectively. At the end of the study, the daily dose will be decreased by 250 mg/month rate.
  Other Names: Nicotinic acid

SUMMARY:
The most frequent form of adult-onset mitochondrial disorders is mitochondrial myopathy, often manifesting with progressive external ophthalmoplegia (PEO), progressive muscle weakness and exercise intolerance. Mitochondrial myopathy is often caused by single heteroplasmic mitochondrial DNA (mtDNA) deletions or multiple mtDNA deletions, the former being sporadic and latter caused by mutations in nuclear-encoded proteins of mtDNA maintenance. Currently, no curative treatment exists for this disease. The investigators have previously observed that supplementation with an NAD+ precursor vitamin B3, nicotinamide riboside, prevented and delayed disease symptoms by increasing mitochondrial biogenesis in a mouse model for mitochondrial myopathy. Vitamin B3 exists in several forms: nicotinic acid (niacin), nicotinamide, and nicotinamide riboside, and it has been demonstrated to give power to diseased mitochondria in animal studies by increasing intracellular levels of NAD+, the important cofactor required for the cellular energy metabolism.

In this study, the form of vitamin B3, niacin, was used to activate dysfunctional mitochondria and to rescue signs of mitochondrial myopathy. Of the vitamin B3 forms, niacin, is employed, because it has been used in large doses to treat hypercholesterolemia patients, and has a proven safety record in humans. Phenotypically similar mitochondrial myopathy patients are studied, as the investigator's previous expertise indicates that similar presenting phenotypes predict uniform physiological and clinical responses to interventions, despite varying genetic backgrounds. Patients either with sporadic single mtDNA deletions or a mutation in a Twinkle gene causing multiple mtDNA deletions were recruited. In addition, for every patient, two gender- and age-matched healthy controls are recruited. Clinical examinations and collection of muscle biopsies are performed at the time points 0, 4 and 10 months (patients) or at 0 and 4 months (controls). Fasting blood samples are collected every second week until 4 months and thereafter every six weeks until the end of the study. The effects of niacin on disease markers, muscle mitochondrial biogenesis, muscle strength and the metabolism of the whole body are studied in patients and healthy controls.

The hypothesis is that an NAD+ precursor, niacin, will increase intracellular NAD+ levels, improve mitochondrial biogenesis and alleviate the symptoms of mitochondrial myopathy in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Manifestation of pure mitochondrial myopathy, with no major other symptoms or manifestations, caused by single or multiple deletions of mtDNA
2. Age and gender matched healthy controls for every patient
3. Agreed to avoid vitamin supplementation or nutritional products with vitamin B3 forms 14 days prior to the enrollment and during the study
4. Written, informed consent to participate in the study

Exclusion Criteria:

1. Inability to follow study protocol
2. Pregnancy or breast-feeding at any time of the trial
3. Malignancy that requires continuous treatment
4. Unstable heart disease
5. Severe kidney disease requiring treatment
6. Severe encephalopathy
7. Regular usage of intoxicants

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
NAD+ and related metabolite levels in blood and muscle | Baseline, 4 months and 10 months
  Change in concentrations of NAD+ and related metabolites such as: nicotinamide adenine dinucleotide phosphate, nicotinic acid adenine dinucleotide, nicotinamide, and nicotinamide mononucleotide measured using high performance liquid chromatography-mass spectrometry

SECONDARY OUTCOMES:
Number of diseased muscle fibers | Baseline, 4 months and 10 months
  Change in number of abnormal muscle fibers (frozen sections, in situ histochemical activity analysis of cytochrome c oxidase negative / succinate-dehydrogenase positive muscle fibers; and immunohistochemistry of complex I negative muscle fibers
Mitochondrial biogenesis | Baseline, 4 months and 10 months
  Change in mitochondria immunohistochemical staining intensity
Muscle mitochondrial oxidative capacity | Baseline, 4 months and 10 months
  Change in muscle histochemical activity of mitochondrial cytochrome c oxidase
Muscle metabolomic profile | Baseline, 4 months and 10 months
  Change in muscle metabolite concentrations measured with mass spectrometry
Core muscle strength | Baseline, 4 months and 10 months
  Change in core muscle strength measured by static and dynamic back and abdominal strength tests (number of repeats)
Circulating levels of disease biomarkers, fibroblast growth factor 21 (FGF21) and growth/differentiation factor 15 (GDF15) | Baseline, 4 months and 10 months
  Change in circulating FGF21 and GDF15 concentrations measured using ELISA kits
Muscle mitochondrial DNA deletions | Baseline, 4 months and 10 months
  Change in muscle mtDNA deletion load detected using polymerase chain reaction amplification
Muscle transcriptomic profile | Baseline, 4 months and 10 months
  Change in muscle gene expression determined using RNA sequencing approach

OTHER OUTCOMES:
Body weight and body composition | Baseline, 4 months and 10 months
  Change in body weight as well as fat mass and fat free mass measured with bioimpedance
Ectopic lipid accumulation, i.e. liver and muscle lipid content | Baseline, 4 months and 10 months
  Change in liver and muscle fat content measured with proton magnetic resonance spectroscopy
Circulating lipid profiles | Baseline, 4 months and 10 months
  Change in circulating HDL, LDL and triglyceride concentrations measured using standard photometric enzymatic assay

CONTACTS AND LOCATIONS:
Overall Officials: Anu Suomalainen Wartiovaara, MD,PhD, Principal Investigator — Research Programs Unit, University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suomalainen A, Battersby BJ. Mitochondrial diseases: the contribution of organelle stress responses to pathology. Nat Rev Mol Cell Biol. 2018 Feb;19(2):77-92. doi: 10.1038/nrm.2017.66. Epub 2017 Aug 9. PMID 28792006
- [Background] Ylikallio E, Suomalainen A. Mechanisms of mitochondrial diseases. Ann Med. 2012 Feb;44(1):41-59. doi: 10.3109/07853890.2011.598547. Epub 2011 Aug 2. PMID 21806499
- [Background] Rajman L, Chwalek K, Sinclair DA. Therapeutic Potential of NAD-Boosting Molecules: The In Vivo Evidence. Cell Metab. 2018 Mar 6;27(3):529-547. doi: 10.1016/j.cmet.2018.02.011. PMID 29514064
- [Background] Khan NA, Auranen M, Paetau I, Pirinen E, Euro L, Forsstrom S, Pasila L, Velagapudi V, Carroll CJ, Auwerx J, Suomalainen A. Effective treatment of mitochondrial myopathy by nicotinamide riboside, a vitamin B3. EMBO Mol Med. 2014 Jun;6(6):721-31. doi: 10.1002/emmm.201403943. PMID 24711540
- [Background] Cerutti R, Pirinen E, Lamperti C, Marchet S, Sauve AA, Li W, Leoni V, Schon EA, Dantzer F, Auwerx J, Viscomi C, Zeviani M. NAD(+)-dependent activation of Sirt1 corrects the phenotype in a mouse model of mitochondrial disease. Cell Metab. 2014 Jun 3;19(6):1042-9. doi: 10.1016/j.cmet.2014.04.001. Epub 2014 May 8. PMID 24814483
- [Background] Guyton JR, Bays HE. Safety considerations with niacin therapy. Am J Cardiol. 2007 Mar 19;99(6A):22C-31C. doi: 10.1016/j.amjcard.2006.11.018. Epub 2006 Nov 28. PMID 17368274
- [Background] Vosper H. Niacin: a re-emerging pharmaceutical for the treatment of dyslipidaemia. Br J Pharmacol. 2009 Sep;158(2):429-41. doi: 10.1111/j.1476-5381.2009.00349.x. Epub 2009 Jul 20. PMID 19627285
- [Background] Ahola S, Auranen M, Isohanni P, Niemisalo S, Urho N, Buzkova J, Velagapudi V, Lundbom N, Hakkarainen A, Muurinen T, Piirila P, Pietilainen KH, Suomalainen A. Modified Atkins diet induces subacute selective ragged-red-fiber lysis in mitochondrial myopathy patients. EMBO Mol Med. 2016 Nov 2;8(11):1234-1247. doi: 10.15252/emmm.201606592. Print 2016 Nov. PMID 27647878
- [Background] Suomalainen A, Elo JM, Pietilainen KH, Hakonen AH, Sevastianova K, Korpela M, Isohanni P, Marjavaara SK, Tyni T, Kiuru-Enari S, Pihko H, Darin N, Ounap K, Kluijtmans LA, Paetau A, Buzkova J, Bindoff LA, Annunen-Rasila J, Uusimaa J, Rissanen A, Yki-Jarvinen H, Hirano M, Tulinius M, Smeitink J, Tyynismaa H. FGF-21 as a biomarker for muscle-manifesting mitochondrial respiratory chain deficiencies: a diagnostic study. Lancet Neurol. 2011 Sep;10(9):806-18. doi: 10.1016/S1474-4422(11)70155-7. Epub 2011 Aug 3. PMID 21820356
- [Background] Nikkanen J, Forsstrom S, Euro L, Paetau I, Kohnz RA, Wang L, Chilov D, Viinamaki J, Roivainen A, Marjamaki P, Liljenback H, Ahola S, Buzkova J, Terzioglu M, Khan NA, Pirnes-Karhu S, Paetau A, Lonnqvist T, Sajantila A, Isohanni P, Tyynismaa H, Nomura DK, Battersby BJ, Velagapudi V, Carroll CJ, Suomalainen A. Mitochondrial DNA Replication Defects Disturb Cellular dNTP Pools and Remodel One-Carbon Metabolism. Cell Metab. 2016 Apr 12;23(4):635-48. doi: 10.1016/j.cmet.2016.01.019. Epub 2016 Feb 25. PMID 26924217
- [Background] Khan NA, Nikkanen J, Yatsuga S, Jackson C, Wang L, Pradhan S, Kivela R, Pessia A, Velagapudi V, Suomalainen A. mTORC1 Regulates Mitochondrial Integrated Stress Response and Mitochondrial Myopathy Progression. Cell Metab. 2017 Aug 1;26(2):419-428.e5. doi: 10.1016/j.cmet.2017.07.007. PMID 28768179
- [Derived] Pirinen E, Auranen M, Khan NA, Brilhante V, Urho N, Pessia A, Hakkarainen A, Kuula J, Heinonen U, Schmidt MS, Haimilahti K, Piirila P, Lundbom N, Taskinen MR, Brenner C, Velagapudi V, Pietilainen KH, Suomalainen A. Niacin Cures Systemic NAD+ Deficiency and Improves Muscle Performance in Adult-Onset Mitochondrial Myopathy. Cell Metab. 2020 Jun 2;31(6):1078-1090.e5. doi: 10.1016/j.cmet.2020.04.008. Epub 2020 May 7. PMID 32386566